CLINICAL TRIAL: NCT00219427
Title: Multicenter Clinical Trials of Retina Projection System
Brief Title: Retina Projection System Trials for Low Vision People
Status: Completed | Type: Observational
Sponsor: Osaka City University (Other)
Collaborators: Nihon University (Other); Kurume University (Other); Miyata Eye Hospital (Unknown); Fukuoka Kinen Hospital (Unknown); Kimura Eye and Internal Medicine Hospital (Other)
Responsible Party: Kunihiko Shiraki, MD, Osaka City University, Dept of Ophthalmology
Other Study IDs: OCUM2004681; OCUM2004681
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2008-05-22 (Estimated); Status verified 2008-05

CONDITIONS: Vision, Low
Keywords: Low vision
MeSH Terms: conditions — Vision, Low

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1

SUMMARY:
1. Purpose

   a. Examination on Efficacy of Retina Projection System
2. Patients

   a. Low vision patients
3. Methods

   1. Vision aids

      * Retina Projection System
      * Face-mounted video display as control
   2. Comparison of Reading Speeds with both vision aids

DETAILED DESCRIPTION:
1. Purpose

   a. Examination on efficacy of a new vision aid of Retina Projection System
2. Patients

   1. Low vision patients
   2. Vision between 0.06 and 0.3
   3. no exclusion on kinds of ocular diseases
3. Methods

   1. Vision aids

      * Retina Projection System
      * Face-mounted video display as control
   2. Computer-aided measurement of reading speeds of individual characters
   3. Comparison of reading Speeds with the two vision aids

ELIGIBILITY:
Inclusion Criteria:

* low vision patients
* vision between 0.06 and 0.3

Exclusion Criteria:

* light perception
* hand motion
* vision less than 0.06

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2005-01; Primary Completion 2005-11 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Reading speeds with two different vision aids | Visits for measuring reading speeds

CONTACTS AND LOCATIONS:
Overall Officials: Kunihiko Shiraki, MD, Study Director — Dept. of Ophthalmology and Visual Sciences, Osaka City University, Graduate School of Medicine
Locations (6):
- Japan (6):
  - Fukuoka Kinen Hospital, Fukuoka, Fukuoka
  - Kurume University, Kurume, Fukuoka
  - Kimura Eye and Medical Hospital, Kure, Hiroshima
  - Miyata Eye Hospital, Miyakonojō, Miyazaki
  - Osaka City University, Osaka, Osaka
  - Nihon University Surugadai Hospital, Tokyo, Tokyo